CLINICAL TRIAL: NCT01831037
Title: The Regression of Liver Fibrosis and Risk for Hepatocellular Carcinoma (ROLFH) Study
Acronym: ROLFH
Status: Withdrawn | Type: Observational
Why Stopped: Unable to obtain funding
Sponsor: University of Arkansas (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Toronto (Other); University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: 137855
Record Dates: First submitted 2013-04-02; First posted 2013-04-15 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Hepatitis C; Chronic Hepatitis B
Keywords: Hepatocellular carcinoma; Regressed cirrhosis; Hepatitis C; Hepatitis B; Noninvasive markers of fibrosis; FibroTest; FibroSure; FibroScan; Transient elastography
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis B, Chronic; Carcinoma, Hepatocellular; Hepatitis C; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, PBMC for DNA isolation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Regression of fibrosis: Group conformed by patients experiencing improvement in the noninvasive markers of fibrosis, Fibrotest/Fibrosure and transient elastography, while enrolled in the study.
  Interventions: Other: Regression of fibrosis; Other: Specific risk factors related to hepatocellular carcinoma
- No regression of fibrosis: Group conformed by patients not showing the predefined improvement in the noninvasive markers of fibrosis, Fibrotest/Fibrosure and transient elastography, while enrolled in the study.

INTERVENTIONS:
Other: Regression of fibrosis — Regression of fibrosis will be defined by assessing yearly evolution of noninvasive markers in patients who received antiviral therapy before start of the study, and by comparing baseline markers before start of antiviral therapy to those on subsequent yearly visits in patients prospective recruited (>50% of cases).
  Other Names: FibroTest, FibroSure, FibroScan (transient elastography)
  Groups: Regression of fibrosis
Other: Specific risk factors related to hepatocellular carcinoma — Such as: family history of liver cancer; body mass index; alcohol, smoking and recreational drug use status; dietary habits, including use of caffeinated drinks; comorbidities such as type 2 diabetes mellitus; use of medications for other chronic diseases such as statins and angiotensin-converting enzyme inhibitors.
  Groups: Regression of fibrosis

SUMMARY:
This study aims to demonstrate that patients with chronic hepatitis C (CHC) and B (CHB) experiencing regression of liver cirrhosis after effective antiviral therapy have decreased risk for hepatocellular carcinoma (HCC). Primary aim is to determine the incidence of HCC in patients with cirrhosis secondary to CHC and CHB, after treatment is provided, and to identify the magnitude of the decreased risk for HCC in patients experiencing regression of fibrosis. As a secondary aim, environmental risk factors for HCC development will be sought, in order to determine a subset of patients in whom it will be safe to stop surveillance.

DETAILED DESCRIPTION:
Cirrhosis is the final pathway of chronic liver disease, and up to 30% of patients develop hepatocellular carcinoma (HCC) within 5 years of diagnosis of cirrhosis. Worldwide, chronic hepatitis C (CHC) and B (CHB) account for the majority of cases of cirrhosis. Successful antiviral treatment results in regression of fibrosis in the majority of patients. Surveillance programs for early detection of HCC mandate the use of imaging (ultrasound/CT-scan) every 6 months. It has been shown in CHC and CHB that the risk of HCC is greatly reduced after viral disease is eradicated/inactive. However, the impact that regression of fibrosis and other factors could have in abating the incidence of HCC has not been systematically investigated. Currently, all patients with eradicated/inactive viral disease continue to be enrolled in HCC surveillance programs, generating anxiety in patients and very high costs to our healthcare system. Fibrotest (FT) and transient elastography (TE) are noninvasive tools proven to be useful for serial assessment of liver fibrosis.

OBJECTIVES: The proposed hypothesis is that patients with regression of liver fibrosis have decreased risk for HCC. Primary aim is to determine the incidence of HCC in patients with cirrhosis secondary to CHC and CHB, during the 3-7 years after treatment is provided, and to identify the magnitude of the decreased risk for HCC in patients experiencing regression of fibrosis. As a secondary aim, environmental risk factors for HCC development will be sought, in order to determine a subset of patients in whom it will be safe to stop surveillance.

METHODS: Patients 18-70 year-old with cirrhosis will be identified from hepatology clinics in 4 academic centers in North America. FT/TE will be obtained before the start of antivirals and yearly thereafter (prospective arm). A retrolective arm of all patients treated no earlier than Jan/2009 will also be included. In this group, baseline FT/TE will be performed off treatment (CHC) or after initial phase of therapy (CHB), and yearly thereafter. During baseline and yearly visits other factors possibly affecting HCC development will be investigated (family history, comorbidities, BMI, diet, etc.). Patients will be classified as having or having not undergone regression of fibrosis after a 3-year follow up, depending on FT and TE evolution. During follow up, all patients will undergo 6-month imaging as part of their routine HCC surveillance. Based on power calculations, enrollment should stop after 924 patients have been recruited. Kaplan-Meier and Cox regression models will be used to analyze data.

PATIENT OUTCOMES: ROLFH study uses state-of-the-art noninvasive markers of liver fibrosis to test whether reversed fibrosis decreases the risk of HCC. We believe this study will lead to a better understanding of HCC risk factors, improved patient counseling and decision making, optimized screening and allocation of health resources, and decreased healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Chronic liver disease due to CHC or CHB.
* Starting of disease-specific treatment no earlier than January of 2010. Treatment could consist of:

  * combination therapy with peginterferon and ribavirin, with or without a direct-acting viral agent in CHC;
  * single or combination therapy containing peginterferon, entecavir, or tenofovir in CHB.
* Established cirrhosis on liver biopsy (METAVIR F4) obtained before starting disease-specific treatment.
* In patients without liver biopsy, any of the following criteria will be used as a surrogate to define cirrhosis:

  * History of spleen >13 cm, bilirubin >2, albumin <3.5, INR >1.5 (2 of 3 criteria).
  * History of APRI ([AST/ULN]/platelets x 100) >2, and esophageal varices or ascites.
  * History of Fibrotest/Fibrosure >0.74, and TE >12.5 kPa (M-probe) or >10 kPa (XL-probe).

Exclusion Criteria:

* Known diagnosis of hepatocellular carcinoma or portal vein thrombosis
* Conditions limiting Fibrotest/Fibrosure read: hemolysis, Gilbert's syndrome, autoimmune disease.
* Conditions limiting TE read: ascites, heart failure with retrograde vascular congestion, extrahepatic cholestasis.
* Pregnancy or implantable active medical device (such as pacemaker or defibrillator).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C or B, with cirrhosis, with successful antiviral treatment no earlier than January 2010 (retrospective component), or planned to start antiviral treatment by the time of recruitment
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular carcinoma | 3 years
  According to standard imaging surveillance protocol, and confirmatory CT/MRI/biopsy

SECONDARY OUTCOMES:
Risk factors for hepatocellular carcinoma | Change from baseline to 3 years
  Positive family history of liver cancer, BMI, active/previous smoking, active/previous alcohol consumption, caffeine consumption in diet, diabetes mellitus, use of drugs for chronic medical conditions
Profile with lowest risk for hepatocellular carcinoma | Change from baseline to 3 years
  Composite of regression of fibrosis plus other specific conditions decreasing incidence of hepatocellular carcinoma to <1.5% / year

OTHER OUTCOMES:
Regression of liver fibrosis | Change from baseline to 3 years
  According to Fibrotest/Fibrosure and transient elastography

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duarte-Rojo, MD, MSc, Principal Investigator — University of Arkansas; Jonathan A Dranoff, MD, Principal Investigator — University of Arkansas
Locations (4):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Toronto, Toronto, Ontario

REFERENCES:
- [Background] El-Serag HB. Epidemiology of viral hepatitis and hepatocellular carcinoma. Gastroenterology. 2012 May;142(6):1264-1273.e1. doi: 10.1053/j.gastro.2011.12.061. PMID 22537432
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] Barritt AS 4th, Fried MW. Maximizing opportunities and avoiding mistakes in triple therapy for hepatitis C virus. Gastroenterology. 2012 May;142(6):1314-1323.e1. doi: 10.1053/j.gastro.2012.02.013. PMID 22537438
- [Background] van der Meer AJ, Veldt BJ, Feld JJ, Wedemeyer H, Dufour JF, Lammert F, Duarte-Rojo A, Heathcote EJ, Manns MP, Kuske L, Zeuzem S, Hofmann WP, de Knegt RJ, Hansen BE, Janssen HL. Association between sustained virological response and all-cause mortality among patients with chronic hepatitis C and advanced hepatic fibrosis. JAMA. 2012 Dec 26;308(24):2584-93. doi: 10.1001/jama.2012.144878. PMID 23268517
- [Background] Duarte-Rojo A, Altamirano JT, Feld JJ. Noninvasive markers of fibrosis: key concepts for improving accuracy in daily clinical practice. Ann Hepatol. 2012 Jul-Aug;11(4):426-39. PMID 22700624
- [Background] Myers RP, Pomier-Layrargues G, Kirsch R, Pollett A, Duarte-Rojo A, Wong D, Beaton M, Levstik M, Crotty P, Elkashab M. Feasibility and diagnostic performance of the FibroScan XL probe for liver stiffness measurement in overweight and obese patients. Hepatology. 2012 Jan;55(1):199-208. doi: 10.1002/hep.24624. Epub 2011 Nov 18. PMID 21898479
- [Background] Myers RP, Pomier-Layrargues G, Kirsch R, Pollett A, Beaton M, Levstik M, Duarte-Rojo A, Wong D, Crotty P, Elkashab M. Discordance in fibrosis staging between liver biopsy and transient elastography using the FibroScan XL probe. J Hepatol. 2012 Mar;56(3):564-70. doi: 10.1016/j.jhep.2011.10.007. Epub 2011 Oct 23. PMID 22027584